CLINICAL TRIAL: NCT02365597
Title: A Phase 2, Two-arm Multicenter, Open-Label Study to Determine the Efficacy and the Safety of Two Different Dose Regimens of a Pan-FGFR Tyrosine Kinase Inhibitor JNJ-42756493 in Subjects With Metastatic or Surgically Unresectable Urothelial Cancer With FGFR Genomic Alterations
Brief Title: An Efficacy and Safety Study of Erdafitinib (JNJ-42756493) in Participants With Urothelial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR105065; 42756493BLC2001 (Other: Janssen Research & Development, LLC); 2014-002408-26 (EudraCT Number); 2023-510273-34-00 (Registry Identifier: EUCT number)
Expanded Access: NCT03825484 (Approved for marketing)
Record Dates: First submitted 2015-01-29; First posted 2015-02-19 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Cancer
Keywords: Urothelial Cancer; JNJ-42756493; Erdafitinib; Tyrosine Kinase Inhibitor
MeSH Terms: interventions — erdafitinib; Midazolam; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Erdafitinib (8 milligram) (Experimental): Prior to interim analysis 1 (IA1), there were 2 treatment regimens: Regimen 1 (10 milligram [mg] once daily, 7 days on/7 days off); and Regimen 2 (6 mg once daily for 28 days). Following IA1, Regimen 1 is closed for further enrollment and starting dose of Regimen 2 is increased to 8 mg once daily for 28 days on a 28-day cycle (referred to as Regimen 3). Participants who enrolled in DDI substudy will receive pretreatment with single doses of midazolam (Day -2) and metformin (Day -1). Participants enrolled in DDI substudy will receive 8 mg erdafitinib treatment from Day 1 to Day 15, single doses of midazolam 2.5 mg (Day 13) and metformin 1000 mg (Day 14) and erdafitinib treatment will continued until disease progression. Participants who completed the DDI substudy and continue to benefit from erdafitinib treatment, will continue to receive erdafitinib in long-term extension (LTE) phase.
  Interventions: Drug: Erdafitinib; Drug: Midazolam; Drug: Metformin

INTERVENTIONS:
Drug: Erdafitinib — 8 mg orally once daily for 28 days on a 28 day cycle.
  Other Names: JNJ-42756493
Drug: Midazolam — Participants who enrolled in DDI substudy will receive pretreatment with single dose of midazolam on Day -2 and single dose of midazolam on Day 13.
Drug: Metformin — Participants who enrolled in DDI substudy will receive pretreatment with single dose of metformin on Day -1 and single dose of metformin on Day 14.

SUMMARY:
The purpose of this study is to evaluate the objective response rate (complete response [CR]+ partial response [PR]) of the selected dose regimen in participants with metastatic or surgically unresectable urothelial cancers that harbor specific FGFR genomic alterations.

DETAILED DESCRIPTION:
This is a multicenter, open-label study (participants will know the identity of study drugs administered) to evaluate the efficacy and safety of erdafitinib in participants with urothelial cancer. The study comprises a 30-days Screening Phase, a Treatment Phase comprised of 28-day treatment cycles that will continue until disease progression or unacceptable toxicity occurs in a long-term extension (LTE) phase, and a post-treatment Follow-up Phase that will extend from the End-of-Treatment Visit until the participant has died, withdraws consent, is lost to follow-up, or the end of the study, whichever comes first. The end of study is defined as the date when all participants have completed the study treatment (Regimens 1 to 3) and all participants enrolled under the drug-drug interaction (DDI) substudy are no longer receiving treatment with erdafitinib. The purpose of DDI sub-study is to evaluate the interaction of repeated doses of erdafitinib with a sensitive cytochrome 450 (CYP) 3A substrate (midazolam) and with an organic cation transporter 2 (OCT2) probe substrate (metformin). Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologic demonstration of metastatic or surgically unresectable urothelial cancer. Minor components of variant histology such as glandular or squamous differentiation, or evolution to more aggressive phenotypes such as sarcomatoid or micropapillary change are acceptable
* Must have measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) at baseline
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status score 0, 1, or 2
* Must have adequate bone marrow, liver, and renal function as described in protocol
* Negative pregnancy test (urine or serum beta human chorionic gonadotropin [b-hCG]) at Screening for women of child bearing potential who are sexually active
* Must have shown disease progression according to RECIST, version 1.1, following prior chemotherapy for metastatic or surgically unresectable urothelial cancer. Participants who received neoadjuvant or adjuvant chemotherapy and showed disease recurrence or progression according to RECIST, version 1.1, within 12 months of the last dose are considered to have received chemotherapy in the metastatic setting. These participants will be referred to as chemo-refractory participants. (Participants who have shown disease progression according to RECIST, version 1.1 following prior treatment with anti-Programmed death-ligand 1 (anti PDL1/PD1) antibodies are also eligible) For DDI substudy
* Disease progression following prior chemotherapy for metastatic or surgically unresectable urothelial cancer. Participants who received neoadjuvant or adjuvant chemotherapy and showed disease recurrence or progression within 12 months of the last dose are considered to have received chemotherapy in the metastatic setting

Exclusion Criteria:

* Received chemotherapy, targeted therapies, definitive radiotherapy, or treatment with an investigational anticancer agent within 2 weeks (in the case of nitrosoureas and mitomycin C, within 6 weeks; in the case of immunotherapy, within 4 weeks) before the first administration of study drug. Localized palliative radiation therapy (but should not include radiation to target lesions) and ongoing bisphosphonates and denosumab, are permitted
* Has persistent phosphate level greater than upper limit of normal (ULN) during screening (within 14 days of treatment and prior to Cycle 1 Day 1) and despite medical management
* Has a history of or current uncontrolled cardiovascular disease
* Females who are pregnant, breast-feeding, or planning to become pregnant within 3 months after the last dose of study drug and males ho plan to father a child while enrolled in this study or within 5 months after the last dose of study drug
* Has not recovered from reversible toxicity of prior anticancer therapy (except toxicities which are not clinically significant such as alopecia, skin discoloration, or Grade 1 neuropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2027-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (105):
- United States (25):
  - Sedona, Arizona
  - Los Angeles, California
  - Orange, California
  - Sacramento, California
  - Stanford, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Minneapolis, Minnesota
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - New York, New York
  - Charlotte, North Carolina
  - Medford, Oregon
  - Tualatin, Oregon
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Denton, Texas
  - Houston, Texas
  - Hampton, Virginia
- Austria (3):
  - Graz
  - Linz
  - Vienna
- Belgium (5):
  - Aalst
  - Brussels
  - Charleroi
  - Ghent
  - Wilrijk
- France (11):
  - Angers
  - Bordeaux
  - Caen Cédex 05
  - Dijon
  - Lyon
  - Nice
  - Nîmes
  - Paris
  - Saint-Herblain
  - Suresnes
  - Villejuif
- Germany (14):
  - Berlin
  - Erlangen
  - Essen
  - Freiburg im Breisgau
  - Göttingen
  - Greifswald
  - Hamburg
  - Hanover
  - Heidelberg
  - München
  - Münster
  - Regensburg
  - Straubing
  - Weiden/Opf
- India (4):
  - Bangalore
  - Kolkata
  - Mira Road (East)
  - Nadiād
- Israel (6):
  - Beer Yaakov
  - Beersheba
  - Haifa
  - Kfar Saba
  - Petah Tikva
  - Tel Aviv
- Chisinau, Moldova
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Iași
- Russia (6):
  - Barnaul
  - Moscow
  - Omsk
  - Pyatigorsk
  - Saint Petersburg
  - Ufa
- South Korea (4):
  - Daejeon
  - Goyang-si
  - Incheon
  - Seoul
- Spain (10):
  - Badalona
  - Barcelona
  - Madrid
  - Málaga
  - Pamplona
  - Sabadell
  - Santander
  - Santiago de Compostela
  - Seville
  - Valencia
- Taiwan (4):
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Istanbul, Turkey (Türkiye)
- United Kingdom (7):
  - Blackburn
  - Dundee
  - Essex
  - London
  - Metropolitan Borough of Wirral
  - Plymouth
  - Sutton

REFERENCES:
- [Derived] Siefker-Radtke AO, Necchi A, Park SH, Garcia-Donas J, Huddart RA, Burgess EF, Fleming MT, Rezazadeh Kalebasty A, Mellado B, Varlamov S, Joshi M, Duran I, Tagawa ST, Zakharia Y, Akapame S, Santiago-Walker AE, Monga M, O'Hagan A, Loriot Y; BLC2001 Study Group. Efficacy and safety of erdafitinib in patients with locally advanced or metastatic urothelial carcinoma: long-term follow-up of a phase 2 study. Lancet Oncol. 2022 Feb;23(2):248-258. doi: 10.1016/S1470-2045(21)00660-4. Epub 2022 Jan 11. PMID 35030333
- [Derived] Dosne AG, Valade E, Goeyvaerts N, De Porre P, Avadhani A, O'Hagan A, Li LY, Ouellet D, Perez Ruixo JJ. Exposure-response analyses of erdafitinib in patients with locally advanced or metastatic urothelial carcinoma. Cancer Chemother Pharmacol. 2022 Feb;89(2):151-164. doi: 10.1007/s00280-021-04381-4. Epub 2022 Jan 3. PMID 34977972
- [Derived] Loriot Y, Necchi A, Park SH, Garcia-Donas J, Huddart R, Burgess E, Fleming M, Rezazadeh A, Mellado B, Varlamov S, Joshi M, Duran I, Tagawa ST, Zakharia Y, Zhong B, Stuyckens K, Santiago-Walker A, De Porre P, O'Hagan A, Avadhani A, Siefker-Radtke AO; BLC2001 Study Group. Erdafitinib in Locally Advanced or Metastatic Urothelial Carcinoma. N Engl J Med. 2019 Jul 25;381(4):338-348. doi: 10.1056/NEJMoa1817323. PMID 31340094

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg: Participants received single dose of erdafitinib 10 mg tablet, orally, once daily, starting from Day 1 through Day 7 and from Day 15 through Day 21 and so on, that is 7-day on and off in each subsequent 28-day cycles starting from Cycle 1. Based on serum phosphate (PO4) levels, there was an option to up-titrate erdafitinib dose to 12 mg, orally, once daily starting from Cycle 2 Day 1 until disease progression, unacceptable toxicity, or any other reason for treatment discontinuation.
- Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg: Participants received single dose of erdafitinib 6 mg tablet, orally, once daily, starting from Day 1 through Day 28 in each subsequent 28-day cycles starting from Cycle 1. Based on serum PO4 levels, there was an option to up-titrate erdafitinib dose to 8 mg, orally, once daily starting from Cycle 2 Day 1 until disease progression, unacceptable toxicity, or any other reason for treatment discontinuation.
- Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg: Participants received single dose of erdafitinib 8 mg tablet, orally, once daily, starting from Day 1 through Day 28 in each subsequent 28-day cycles starting from Cycle 1. Based on serum PO4 levels, there was an option to up-titrate erdafitinib dose to 9 mg, orally, once daily starting from Cycle 1 Day 15 until disease progression, unacceptable toxicity, or any other reason for treatment discontinuation.
- Drug-Drug Interaction (DDI) Sub-study: Midazolam 2.5 mg + Metformin 1000 mg + Erdafitinib 8/9 mg: Participants received pretreatment with single doses of midazolam 2.5 mg syrup orally on Day -2 and metformin 1000 mg tablet orally on Day -1 along with erdafitinib 8 mg tablet, orally, on 28-day cycles starting from Cycle 1 Day 1 to Day 15 (or up-titrated to 9 mg on Day 15 based on Day 14 serum PO4 levels) until disease progression, unacceptable toxicity, or any other reason for treatment discontinuation.
Period: Overall Study
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg | Drug-Drug Interaction (DDI) Sub-study: Midazolam 2.5 mg + Metformin 1000 mg + Erdafitinib 8/9 mg
Started | 33 | 79 | 102 | 25
Treated (Safety Analysis Set) | 33 | 78 | 101 | 25
Completed | 31 | 62 | 83 | 6
Not Completed | 2 | 17 | 19 | 19
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 8 | 5 | 1
Not completed — Sponsor's decision | 1 | 3 | 13 | 0
Not completed — Other | 0 | 4 | 0 | 0
Not completed — Enrolled but not treated | 0 | 1 | 1 | 0
Not completed — Ongoing | 0 | 0 | 0 | 17

BASELINE CHARACTERISTICS:
Population: Safety analysis set included participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg | Drug-Drug Interaction (DDI) Sub-study: Midazolam 2.5 mg + Metformin 1000 mg + Erdafitinib 8/9 mg | Total
Number analyzed (Participants) | 33 | 78 | 101 | 25 | 237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 39 | 39 | 11 | 100
  >=65 years | 22 | 39 | 62 | 14 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (7.98) | 64.5 (10.36) | 66.1 (10.2) | 64.8 (10.35) | 65.8 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 24 | 24 | 10 | 69
  Male | 22 | 54 | 77 | 15 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 1 | 6
  Not Hispanic or Latino | 25 | 68 | 75 | 22 | 190
  Unknown or Not Reported | 7 | 8 | 24 | 2 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 11 | 5 | 0 | 18
  Black or African American | 0 | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 24 | 56 | 75 | 20 | 175
  More than one race | 0 | 0 | 0 | 3 | 3
  Unknown or Not Reported | 7 | 7 | 18 | 2 | 34
  Other | 0 | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRIA | 0 | 2 | 2 | 0 | 4
  BELGIUM | 3 | 2 | 4 | 0 | 9
  FRANCE | 7 | 9 | 20 | 1 | 37
  GERMANY | 0 | 5 | 6 | 0 | 11
  INDIA | 0 | 0 | 0 | 3 | 3
  ISRAEL | 0 | 2 | 3 | 0 | 5
  ITALY | 4 | 12 | 19 | 0 | 35
  MOLDOVA, REPUBLIC OF | 0 | 1 | 0 | 0 | 1
  ROMANIA | 0 | 1 | 1 | 0 | 2
  RUSSIAN FEDERATION | 1 | 7 | 11 | 0 | 19
  SOUTH KOREA | 2 | 9 | 3 | 0 | 14
  SPAIN | 7 | 8 | 4 | 20 | 39
  TAIWAN | 0 | 2 | 2 | 0 | 4
  TURKEY | 0 | 0 | 0 | 1 | 1
  UNITED KINGDOM | 1 | 5 | 5 | 0 | 11
  UNITED STATES | 8 | 13 | 21 | 0 | 42

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Percentage of Participants With Best (Overall) Objective Response
Description: Percentage of participants with best (overall) objective response were reported. Best objective response is defined as the best (overall) objective response a participants achieved during the study in the order of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), where CR and PR were confirmed as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. As per RECIST version 1.1, CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in the short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Responders are participants with BOR of CR or PR.
Time Frame: From Cycle 1 Day 1 up to 6 years 2 months
Population: The population included participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 33 | 78 | 101
Percentage of Participants | 21.2 | 34.6 | 39.6

2. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Maximum Observed Plasma Concentration (Cmax) of Midazolam Alone or in Combination With Erdafitinib
Description: Cmax is the maximum observed plasma concentration of midazolam alone or in combination with erdafitinib.
Time Frame: Cycle 1 Day -2 (predose) up to Day 13 post dose
Population: Pharmacokinetic analysis set included all participants who received at least 1 dose of study drug and had at least 1 sample collected during treatment to determine the drug concentration. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- DDI Study: Midazolam 2.5 mg Alone: Participants received single dose of pretreatment midazolam 2.5 mg syrup, orally, once daily, starting from Day -2 through Day 13 of Cycle 1 (each cycle length=28 days).
- DDI Study: Midazolam 2.5 mg + Erdafitinib 8 mg: Participants received single dose of pretreatment midazolam 2.5 mg syrup, orally, once daily, starting from Day -2 through Day 13 of Cycle 1 along with erdafitinib 8 mg starting from Day 1 up to Day 15 of Cycle 1 (each cycle length=28 days).
Arm/Group | DDI Study: Midazolam 2.5 mg Alone | DDI Study: Midazolam 2.5 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 23 | 22
nanograms per milliliter (ng/mL) | 18.4 (7.32) | 15.4 (5.90)

3. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Maximum Observed Plasma Concentration (Cmax) of 1-OH-Midazolam (Midazolam Metabolite) Alone or in Combination With Erdafitinib
Description: Cmax is the maximum observed plasma concentration of 1-OH-Midazolam (midazolam metabolite) alone or in combination with erdafitinib.
Time Frame: Cycle 1 Day -2 (predose) up to Day 13 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- DDI Study: 1-OH-Midazolam 2.5 mg Alone: Participants received single dose of pretreatment 1-OH-Midazolam 2.5 mg syrup, orally, once daily, starting from Day -2 through Day 13 of Cycle 1 (each cycle length=28 days).
- DDI Study: 1-OH-Midazolam 2.5 mg + Erdafitinib 8 mg: Participants received single dose of pretreatment 1-OH-Midazolam 2.5 mg syrup, orally, once daily, starting from Day -2 through Day 13 of Cycle 1 along with erdafitinib 8 mg starting from Day 1 up to Day 15 of Cycle 1 (each cycle length=28 days).
Arm/Group | DDI Study: 1-OH-Midazolam 2.5 mg Alone | DDI Study: 1-OH-Midazolam 2.5 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 23 | 22
ng/mL | 5.39 (3.42) | 4.82 (2.60)

4. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Maximum Observed Plasma Concentration (Cmax) of Metformin Alone or in Combination With Erdafitinib
Description: Cmax is the maximum observed plasma concentration of metformin alone or in combination with erdafitinib
Time Frame: Cycle 1 Day -1 (predose) up to Day 14 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- DDI Study: Metformin 1000 mg Alone: Participants received single dose of metformin 1000 mg tablet, orally, once daily, starting from Day -1 through Day 14 of Cycle 1 (each cycle length=28 days).
- DDI Study: Metformin 1000 mg + Erdafitinib 8 mg: Participants received single dose of metformin 1000 mg tablet, orally, once daily, starting from Day -1 through Day 14 of Cycle 1 along with erdafitinib 8 mg starting from Day 1 up to Day 15 of Cycle 1 (each cycle length=28 days).
Arm/Group | DDI Study: Metformin 1000 mg Alone | DDI Study: Metformin 1000 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 2465 (986) | 2687 (1127)

5. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Midazolam Alone or in Combination With Erdafitinib
Description: Tmax is the time to reach the maximum observed plasma concentration of midazolam alone or in combination with erdafitinib.
Time Frame: Cycle 1 Day -2 (predose) up to Day 13 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | DDI Study: Midazolam 2.5 mg Alone | DDI Study: Midazolam 2.5 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 23 | 22
Hours | 0.50 [0.47 to 1.08] | 0.58 [0.45 to 2.00]

6. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of 1-OH-Midazolam (Midazolam Metabolite) Alone or in Combination With Erdafitinib
Description: Tmax is the time to reach the maximum observed plasma concentration of 1-OH-Midazolam alone or in combination with erdafitinib.
Time Frame: Cycle 1 Day -2 (predose) up to Day 13 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | DDI Study: 1-OH-Midazolam 2.5 mg Alone | DDI Study: 1-OH-Midazolam 2.5 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 23 | 22
Hours | 0.58 [0.47 to 2.08] | 0.58 [0.45 to 4.00]

7. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Metformin Alone or in Combination With Erdafitinib
Description: Tmax is the time to reach maximum observed plasma concentration of metformin alone or in combination with erdafitinib
Time Frame: Cycle 1 Day -1 (predose) up to Day 14 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | DDI Study: Metformin 1000 mg Alone | DDI Study: Metformin 1000 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 20 | 19
Hours | 2.04 [0.42 to 5.00] | 3.00 [0.50 to 8.08]

8. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUC[0-last]) of Midazolam Alone or in Combination With Erdafitinib
Description: AUC(0-last) is the area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration of midazolam alone or in combination with erdafitinib.
Time Frame: Cycle 1 Day -2 (predose) up to Day 13 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Nanograms hours per milliliter (ng*h/mL)
Arm/Group | DDI Study: Midazolam 2.5 mg Alone | DDI Study: Midazolam 2.5 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 23 | 22
Nanograms hours per milliliter (ng*h/mL) | 64.4 (26.8) | 57.1 (27.2)

9. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUC[0-last]) of 1-OH-Midazolam (Midazolam Metabolite) Alone or in Combination With Erdafitinib
Description: AUC(0-last) is the area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration of 1-OH-Midazolam alone or in combination with erdafitinib.
Time Frame: Cycle 1 Day -2 (predose) up to Day 13 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DDI Study: 1-OH-Midazolam 2.5 mg Alone | DDI Study: 1-OH-Midazolam 2.5 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 23 | 22
ng*h/mL | 15.8 (9.59) | 15.1 (10.4)

10. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUC[0-last]) of Metformin Alone or in Combination With Erdafitinib
Description: AUC(0-last) is the area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration of metformin alone or in combination with erdafitinib.
Time Frame: Cycle 1 Day -1 (predose) up to Day 14 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DDI Study: Metformin 1000 mg Alone | DDI Study: Metformin 1000 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 20 | 19
ng*h/mL | 22015 (11967) | 26917 (17973)

11. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Infinite Time (AUC[0-Infinity]) of Midazolam Alone or in Combination With Erdafitinib
Description: AUC(0-Infinity) is the area under the plasma concentration versus time curve from time 0 to the infinite time of midazolam alone or in combination with erdafitinib.
Time Frame: Cycle 1 Day -2 (predose) up to Day 13 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DDI Study: Midazolam 2.5 mg Alone | DDI Study: Midazolam 2.5 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 20 | 17
ng*h/mL | 69.8 (30.5) | 55.9 (28.2)

12. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Infinite Time (AUC[0-Infinity]) of 1-OH-Midazolam (Midazolam Metabolite) Alone or in Combination With Erdafitinib
Description: AUC(0-Infinity) is the area under the plasma concentration versus time curve from time 0 to the infinite time of 1-OH-Midazolam alone or in combination with erdafitinib.
Time Frame: Cycle 1 Day -2 (predose) up to Day 13 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DDI Study: 1-OH-Midazolam 2.5 mg Alone | DDI Study: 1-OH-Midazolam 2.5 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 18 | 13
ng*h/mL | 18.1 (10.8) | 18.4 (13.2)

13. Primary Outcome: Drug-Drug Interaction (DDI) Substudy: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Infinite Time (AUC[0-Infinity]) of Metformin Alone or in Combination With Erdafitinib
Description: AUC(0-Infinity) is the area under the plasma concentration versus time curve from time 0 to the infinite time of metformin alone or in combination with erdafitinib
Time Frame: Cycle 1 Day -1 (predose) up to Day 14 post dose (each cycle length=28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DDI Study: Metformin 1000 mg Alone | DDI Study: Metformin 1000 mg + Erdafitinib 8 mg
Number analyzed (Participants) | 20 | 17
ng*h/mL | 22917 (12539) | 28853 (21738)

14. Secondary Outcome: Main Study: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the duration from the date of the first dose of study drug until the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death due to any cause, whichever occurs first, regardless of the use of subsequent anticancer therapy. As per RECIST version 1.1, CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in the short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From screening up to 6 years 2 months
Population: The population included participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 33 | 78 | 101
months | 4.80 [1.1 to 25.3] | 5.26 [0.4 to 57.9] | 5.52 [0.0 to 51.5]

15. Secondary Outcome: Main Study: Duration of Response (DoR)
Description: DOR is defined as the time (in months) from the date of first observation of response (PR or CR) to the date of the first observation of progression or date of death, whatever the cause based on the RECIST version 1.1. CR: disappearance of all target and non-target lesions. All pathological (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From screening up to 6 years 2 months
Population: The population included participants who received at least 1 dose of study drug and who had CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 7 | 27 | 40
months | 13.37 [4.2 to 19.4] | 4.90 [2.5 to 56.5] | 5.98 [2.4 to 50.2]

16. Secondary Outcome: Main Study: Overall Survival
Description: Overall survival is defined as the time from the date of first dose of study drug to the date of the participant's death from any cause.
Time Frame: From screening up to 6 years 2 months
Population: The population included participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 33 | 78 | 101
months | 7.46 [1.7 to 64.0] | 8.64 [0.4 to 60.1] | 11.30 [0.7 to 56.9]

17. Secondary Outcome: Main Study: Percentage of Participants With Treatment-emergent Adverse Event (TEAEs)
Description: Percentage of participants with TEAEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are those events that occurred from first dose date through 30 days after last dose date, or day before subsequent anticancer therapy, whichever occurs first.
Time Frame: From Day 1 up to 6 years 2 months
Population: The population included participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 33 | 78 | 101
Percentage of Participants | 100 | 100 | 100

18. Secondary Outcome: Main Study: Plasma Concentration of Erdafitinib at 2 Hours (C2h)
Description: C2h is the plasma concentration of erdafitinib at 2 hours.
Time Frame: Cycle 1 Days 1 and 21: Pre-dose up to 2 hours post-dose (each cycle length=28 days)
Population: Pharmacokinetic analysis set included all participants who received at least 1 dose of study drug and had at least 1 sample collected during treatment to determine the drug concentration. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 32 | 74 | 92
ng/mL
  Cycle 1 Day 1 | 529.5 (224.9) | 311.0 (134.8) | 373.0 (168.1)
  Cycle 1 Day 21: number analyzed (Participants) | 23 | 59 | 45
  Cycle 1 Day 21 | 1686.5 (872.3) | 1255.1 (640.0) | 1371.4 (586.6)

19. Secondary Outcome: Main Study: Plasma Concentration of Erdafitinib at 4 Hours (C4h)
Description: C4h is the plasma concentration of erdafitinib at 4 hours.
Time Frame: Cycle 1 Days 1 and 21: Pre-dose up to 4 hours post-dose (each cycle length=28 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg
Number analyzed (Participants) | 32 | 74 | 91
ng/mL
  Cycle 1 Day 1 | 504.0 (189.6) | 290.0 (117.9) | 365.3 (155.6)
  Cycle 1 Day 21: number analyzed (Participants) | 24 | 60 | 46
  Cycle 1 Day 21 | 1753.4 (917.8) | 1257.4 (663.2) | 1329.9 (550.1)

ADVERSE EVENTS:
Time Frame: Main study: From Day 1 up to 6 years 2 months; DDI study: From Day 1 up to 1 year 6 months
Description: The population included participants who received at least 1 dose of study drug.
Arm/Group | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg | Drug-Drug Interaction (DDI) Sub-study: Midazolam 2.5 mg + Metformin 1000 mg + Erdafitinib 8/9 mg
All-Cause Mortality (participants affected / at risk) | 31/33 | 62/78 | 83/101 | 3/25
Serious Adverse Events (participants affected / at risk) | 14/33 | 39/78 | 47/101 | 9/25
Other Adverse Events (participants affected / at risk) | 32/33 | 78/78 | 101/101 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg (N=33) | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg (N=78) | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg (N=101) | Drug-Drug Interaction (DDI) Sub-study: Midazolam 2.5 mg + Metformin 1000 mg + Erdafitinib 8/9 mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angle Closure Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 1 | 2 | 0
Corneal Erosion (Eye disorders) | 0 | 0 | 1 | 0
Detachment of Retinal Pigment Epithelium (Eye disorders) | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 2 | 0
Maculopathy (Eye disorders) | 0 | 0 | 1 | 0
Optic Atrophy (Eye disorders) | 0 | 0 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 1 | 0
Retinal Oedema (Eye disorders) | 0 | 0 | 1 | 0
Retinopathy (Eye disorders) | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1 | 0
Vitreous Detachment (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterocutaneous Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 2 | 0
Breakthrough Pain (General disorders) | 0 | 0 | 1 | 0
Condition Aggravated (General disorders) | 0 | 0 | 1 | 0
Disease Progression (General disorders) | 0 | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 1 | 2 | 2 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0
Performance Status Decreased (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 1 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0 | 0
Eye Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0
Infective Corneal Ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Pelvic Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Periorbital Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 0
Sepsis (Infections and infestations) | 1 | 2 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 4 | 4 | 1
Urosepsis (Infections and infestations) | 0 | 3 | 2 | 0
Bone Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Exposure to Toxic Agent (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Eastern Cooperative Oncology Group Performance Status Worsened (Investigations) | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ureteral Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Brain Oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Mental Impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Device Dislocation (Product Issues) | 1 | 0 | 0 | 0
Device Expulsion (Product Issues) | 0 | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination, Visual (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 3 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephropathy Toxic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 1 | 0
Renal Injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Pain (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Regimen 1: Erdafitinib 10 Milligrams (mg)/ 12 mg (N=33) | Main Study: Regimen 2: Erdafitinib 6 mg/ 8 mg (N=78) | Main Study: Regimen 3: Erdafitinib 8 mg/ 9 mg (N=101) | Drug-Drug Interaction (DDI) Sub-study: Midazolam 2.5 mg + Metformin 1000 mg + Erdafitinib 8/9 mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 8 | 13 | 23 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 6 | 1
Blepharitis (Eye disorders) | 0 | 1 | 6 | 0
Cataract (Eye disorders) | 1 | 4 | 4 | 2
Chorioretinopathy (Eye disorders) | 2 | 2 | 7 | 1
Dry Eye (Eye disorders) | 3 | 7 | 28 | 2
Keratitis (Eye disorders) | 3 | 1 | 4 | 2
Lacrimation Increased (Eye disorders) | 6 | 13 | 12 | 4
Ocular Toxicity (Eye disorders) | 0 | 0 | 0 | 2
Punctate Keratitis (Eye disorders) | 0 | 0 | 5 | 3
Retinal Detachment (Eye disorders) | 1 | 5 | 3 | 3
Vision Blurred (Eye disorders) | 5 | 5 | 18 | 4
Visual Acuity Reduced (Eye disorders) | 0 | 1 | 7 | 1
Visual Impairment (Eye disorders) | 1 | 3 | 7 | 0
Abdominal Pain (Gastrointestinal disorders) | 5 | 14 | 8 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 6 | 9 | 4
Constipation (Gastrointestinal disorders) | 14 | 20 | 29 | 8
Diarrhoea (Gastrointestinal disorders) | 15 | 39 | 56 | 15
Dry Mouth (Gastrointestinal disorders) | 16 | 31 | 46 | 9
Dyspepsia (Gastrointestinal disorders) | 4 | 9 | 12 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 5 | 6 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1 | 7 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 16 | 22 | 4
Stomatitis (Gastrointestinal disorders) | 16 | 34 | 60 | 14
Vomiting (Gastrointestinal disorders) | 8 | 11 | 15 | 1
Asthenia (General disorders) | 10 | 17 | 22 | 9
Chills (General disorders) | 2 | 2 | 2 | 0
Fatigue (General disorders) | 7 | 21 | 33 | 2
Mucosal Dryness (General disorders) | 1 | 1 | 2 | 2
Oedema Peripheral (General disorders) | 5 | 6 | 10 | 1
Pyrexia (General disorders) | 5 | 14 | 13 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 3 | 2
Conjunctivitis (Infections and infestations) | 5 | 7 | 13 | 3
Paronychia (Infections and infestations) | 2 | 12 | 19 | 5
Pneumonia (Infections and infestations) | 1 | 4 | 2 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 10 | 15 | 3
Alanine Aminotransferase Increased (Investigations) | 2 | 9 | 19 | 9
Aspartate Aminotransferase Increased (Investigations) | 3 | 9 | 13 | 9
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 7 | 7 | 2
Blood Creatinine Increased (Investigations) | 5 | 7 | 10 | 2
Weight Decreased (Investigations) | 3 | 8 | 18 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 11 | 28 | 41 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 7 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 4 | 6 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 6 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 16 | 52 | 79 | 19
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3 | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 6 | 13 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 7 | 12 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3 | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 9 | 8 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 12 | 5 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 9 | 14 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 5 | 0
Dysgeusia (Nervous system disorders) | 7 | 7 | 33 | 5
Headache (Nervous system disorders) | 1 | 6 | 7 | 2
Paraesthesia (Nervous system disorders) | 0 | 4 | 3 | 2
Partial Seizures (Nervous system disorders) | 0 | 0 | 0 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 2 | 5 | 4
Taste Disorder (Nervous system disorders) | 3 | 3 | 10 | 0
Tremor (Nervous system disorders) | 2 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 5 | 0
Insomnia (Psychiatric disorders) | 3 | 8 | 9 | 0
Dysuria (Renal and urinary disorders) | 0 | 3 | 6 | 5
Haematuria (Renal and urinary disorders) | 3 | 5 | 11 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 2 | 2
Renal Impairment (Renal and urinary disorders) | 1 | 2 | 8 | 0
Pelvic Pain (Reproductive system and breast disorders) | 2 | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 11 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 7 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 9 | 1
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 9 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 10 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 10 | 34 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 9 | 18 | 34 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 7 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 1 | 7 | 13 | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 4 | 11 | 4
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 2 | 7 | 17 | 9
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 7 | 13 | 19 | 5
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 8 | 7 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 | 14 | 25 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6 | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 7 | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 2 | 1 | 6 | 0
Hypertension (Vascular disorders) | 1 | 0 | 7 | 0
Hypotension (Vascular disorders) | 2 | 6 | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT02365597/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT02365597/SAP_001.pdf